CLINICAL TRIAL: NCT06616441
Title: The Effect of Intraperitoneal Instillation of Bupivacaine on Postoperative Pain After Surgical Laparoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: El Shatby University Hospital for Obstetrics and Gynecology (Other)
Responsible Party: Principal Investigator, Aly Hussein, primary investigator, El Shatby University Hospital for Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0107909
Record Dates: First submitted 2023-12-04; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Grouo A (Active Comparator): Patients that will receive intraoperative instillation of bupivacaine.
  Interventions: Drug: Bupivacaine
- Group B (No Intervention): (Control group) that will not receive the medication.

INTERVENTIONS:
Drug: Bupivacaine — Group (A) only will receive intra-peritoneal 40 ml bupivacaine 0.2%, after laparoscopic procedure before removing trocars.
  Arms: Grouo A

SUMMARY:
Pain after surgical laparoscopy is due to various causes, such as : trocar insertion stimulating somatic pain receptors in the skin ,chemical irritation of peritoneal nerves due to abdominal distension by CO2 which is transformed into carbonic acid in nerves, distention secondary to pneumoperitoneum causes mechanical irritation of visceral and parietal nerves of the peritoneum, furthermore the surgical intervention causing injury and inflammation of the tissues, spillage of blood or serous fluid causing more irritation to the visceral and parietal nerves of the peritoneum which leads to visceral dull aching pain referred mainly to the distribution of the nerve dermatomal area.

Unfortunately, pain is the major complaint of the patients, thus making its evaluation a fundamental requisite in the outcome assessment in our practice. Pain intensity, duration and related disability are the aspects that define pain and its effects. For each of these aspects, different assessment tools exist.

Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' The patient is asked to mark his pain level on the line between the two endpoints.

There are numerous interventions that are associated with reduction in the incidence, severity or both of pain or a reduction in analgesia requirements for women having surgical laparoscopy for gynecological purposes.

Bupivacaine, is a local anesthetic. In nerve blocks, it is injected around the nerve that supplies a certain area, or into the spinal canal's epidural space, bupivacaine binds to the intracellular portion of voltage-gated sodium channels and blocks sodium influx into nerve cells, which prevents depolarization. Without depolarization, no initiation or conduction of a pain signal can occur.

Hence the idea of our study is to instill bupivacaine in a certain concentration in the peritoneal cavity in an attempt to reduce postoperative pain after surgical laparoscopy for gynecological purposes that will inflect certainly on patient's hospital stay and mobility.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted for (80) women undergoing laparoscopic procedures at endoscopy unit at El-Shatby Maternity University Hospital, after approval of ethical committee of Alexandria Faculty of Medicine.

Randomization will be through opaque sealed envelopes.

After signing their informed consents, the patients who are included in the study will be divided into two groups each group include (60) patients.

Group A: Patients that will receive intraoperative instillation of bupivacaine. Group B: (Control group) that will not receive the medication.

The patients in both groups will be subjected to:

Pre-operative:

History taking (gynecological, obstetric, medical any drug reaction and surgical), general examination and abdominal examination.

Intra-operative:

premedication : 1.5 microgram/kg fentanyl IV induction of anathesia: 2mg/kg Propofol IV , 0.5 mg/kg Atracurium IV , ventilation via face mask 2-3 minutes , then endotracheal intubation

1gm paracetamol IV as intraoperative analgesia which will not interfere with postoperative pain scoring.

Group (A) only will receive intra-peritoneal 40 ml bupivacaine 0.2%, after laparoscopic procedure before removing trocars.

ELIGIBILITY:
Inclusion Criteria:

1. Patients those are indicated for surgical laparoscopy, whatever the gynecological problem.
2. Age between (18-50) years.
3. Cooperative patient that can express pain and score it.

Exclusion Criteria:

1. Non-cooperative patients that cannot express and score pain.
2. Drug abusers due to altered pain threshold.
3. Surgical laparoscopy indicated for oncological procedures.
4. Any allergy or reaction to any of the derivatives of bupivacaine drug group.
5. Any cardio-pulmonary condition.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of instilling bupivacaine intraperitoneal in reducing postoperative pain after surgical laparoscopy for gynecologic procedures. | up to 1 day
  Evaluate the efficacy of instilling bupivacaine intraperitoneal in reducing postoperative pain after surgical laparoscopy for gynecologic procedures.

SECONDARY OUTCOMES:
Assessment of the timing passed postoperative, since the patient needs to start the first analgesic dose. | up to 1 day
  Assessment of the timing passed postoperative, since the patient needs to start the first analgesic dose.
Frequency of analgesia requested by the patient in postoperative period. | up to 1 day
  Frequency of analgesia requested by the patient in postoperative period.
Assessment of the time passed postoperative since the patient start mobility | up to 1 day
  Assessment of the time passed postoperative since the patient start mobility

CONTACTS AND LOCATIONS:
Overall Officials: Aly Hussein, Dr, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Cho M, Kim CJ, Hahm TS, Lee YY, Kim TJ, Lee JW, Kim BG, Bae DS, Choi CH. Combination of a pulmonary recruitment maneuver and intraperitoneal bupivacaine for the reduction of postoperative shoulder pain in gynecologic laparoscopy: a randomized, controlled trial. Obstet Gynecol Sci. 2020 Mar;63(2):187-194. doi: 10.5468/ogs.2020.63.2.187. Epub 2020 Feb 20. PMID 32206659
- [Background] Cunningham TK, Draper H, Bexhell H, Allgar V, Allen J, Mikl D, Phillips K. A double-blinded randomised controlled study to investigate the effect of intraperitoneal levobupivacaine on post laparoscopic pain. Facts Views Vis Obgyn. 2020 Oct 8;12(3):155-161. PMID 33123690
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Adlan ASA, Azhary JMK, Tarmidzi HZM, Kamarudin M, Lim RCS, Ng DSW. Post Laparoscopy Pain Reduction Project I (POLYPREP I): intraperitoneal normal saline instillation-a randomised controlled trial. BMC Womens Health. 2022 Apr 12;22(1):116. doi: 10.1186/s12905-022-01696-z. PMID 35413905
- [Background] Sao CH, Chan-Tiopianco M, Chung KC, Chen YJ, Horng HC, Lee WL, Wang PH. Pain after laparoscopic surgery: Focus on shoulder-tip pain after gynecological laparoscopic surgery. J Chin Med Assoc. 2019 Nov;82(11):819-826. doi: 10.1097/JCMA.0000000000000190. PMID 31517775
- [Background] Kaloo P, Armstrong S, Kaloo C, Jordan V. Interventions to reduce shoulder pain following gynaecological laparoscopic procedures. Cochrane Database Syst Rev. 2019 Jan 30;1(1):CD011101. doi: 10.1002/14651858.CD011101.pub2. PMID 30699235
- [Background] Jimenez Cruz J, Diebolder H, Dogan A, Mothes A, Rengsberger M, Hartmann M, Meissner W, Runnebaum IB. Combination of pre-emptive port-site and intraoperative intraperitoneal ropivacaine for reduction of postoperative pain: a prospective cohort study. Eur J Obstet Gynecol Reprod Biol. 2014 Aug;179:11-6. doi: 10.1016/j.ejogrb.2014.05.001. Epub 2014 May 13. PMID 24965972
- [Background] Arden D, Seifert E, Donnellan N, Guido R, Lee T, Mansuria S. Intraperitoneal instillation of bupivacaine for reduction of postoperative pain after laparoscopic hysterectomy: a double-blind randomized controlled trial. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):620-6. doi: 10.1016/j.jmig.2013.03.012. Epub 2013 May 22. PMID 23706546
- [Background] Manjunath AP, Chhabra N, Girija S, Nair S. Pain relief in laparoscopic tubal ligation using intraperitoneal lignocaine: a double masked randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2012 Nov;165(1):110-4. doi: 10.1016/j.ejogrb.2012.06.035. Epub 2012 Jul 21. PMID 22819575
- [Background] Marks JL, Ata B, Tulandi T. Systematic review and metaanalysis of intraperitoneal instillation of local anesthetics for reduction of pain after gynecologic laparoscopy. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):545-53. doi: 10.1016/j.jmig.2012.04.002. Epub 2012 Jul 3. PMID 22763313
- [Background] Malhotra N, Chanana C, Roy KK, Kumar S, Rewari V, Sharma JB. To compare the efficacy of two doses of intraperitoneal bupivacaine for pain relief after operative laparoscopy in gynecology. Arch Gynecol Obstet. 2007 Oct;276(4):323-6. doi: 10.1007/s00404-007-0337-1. Epub 2007 Jul 25. PMID 17653742
- [Background] Chou YJ, Ou YC, Lan KC, Jawan B, Chang SY, Kung FT. Preemptive analgesia installation during gynecologic laparoscopy: a randomized trial. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):330-5. doi: 10.1016/j.jmig.2005.05.005. PMID 16036193
- [Background] Buck L, Varras MN, Miskry T, Ruston J, Magos A. Intraperitoneal bupivacaine for the reduction of postoperative pain following operative laparoscopy: a pilot study and review of the literature. J Obstet Gynaecol. 2004 Jun;24(4):448-51. doi: 10.1080/01443610410001685637. PMID 15203590

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT06616441/SAP_000.pdf